CLINICAL TRIAL: NCT04263168
Title: Glycemic Index Variations In the Early Period Following Bariatric Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Dr. Nir Horesh resident Department of Surgery and Transplant, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6397-19-SMC
Record Dates: First submitted 2019-10-19; First posted 2020-02-10 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus; Bariatric Surgery Candidate
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Bariatric surgery candidates for two types of bariatric surgery, i.e. sleeve gastrectomy (n=80) and Roux-en-Y gastric bypass (RYGB, n=80) will be recruited to the study from the bariatric surgery clinic in the Sheba medical center and will be followed pre- and postoperatively. A control group of candidates for another non-bariatric upper-GI surgery, i.e. cholecystectomy (n=80), will be recruited as well. All participants will undergo medical and metabolic profiling before surgery at baseline, and during the first two weeks following surgery. Metabolic profiling will take place during a run-in session in the Sheba medical center, that will include (A) A detailed briefing on study design, goals, samples collection and OGTT, as well as home sample-collecting kit distribution (B) Installation of a continuous glucose monitoring system (CGM, Abbott 'freeStyle Libre').
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bariatric Surgery Candidates (Experimental): All participants will undergo medical and metabolic profiling before surgery at baseline, and during the first two weeks following surgery. Metabolic profiling will take place during a run-in session in the Sheba medical center, that will include (A) A detailed briefing on study design, goals, samples collection and OGTT, as well as home sample-collecting kit distribution (B) Installation of a continuous glucose monitoring system (CGM, Abbott 'freeStyle Libre').
  Interventions: Diagnostic Test: Continuous Glucose monitoring in the perioperative period
- Laparoscopy Cholecystectomy (Sham Comparator): All participants will undergo medical and metabolic profiling before surgery at baseline, and during the first two weeks following surgery. Metabolic profiling will take place during a run-in session in the Sheba medical center, that will include (A) A detailed briefing on study design, goals, samples collection and OGTT, as well as home sample-collecting kit distribution (B) Installation of a continuous glucose monitoring system (CGM, Abbott 'freeStyle Libre').
  Interventions: Diagnostic Test: Continuous Glucose monitoring in the perioperative period

INTERVENTIONS:
Diagnostic Test: Continuous Glucose monitoring in the perioperative period — All participants will undergo medical and metabolic profiling before surgery at baseline, and during the first two weeks following surgery. Metabolic profiling will take place during a run-in session in the Sheba medical center, that will include (A) A detailed briefing on study design, goals, samples collection and OGTT, as well as home sample-collecting kit distribution (B) Installation of a continuous glucose monitoring system (CGM, Abbott 'freeStyle Libre').

SUMMARY:
The diverse community of gut microbes commonly referred to as the 'gut microbiome', is increasingly suggested to play significant roles in health and disease, and to affect even distant non-GI organs by metabolite signaling. Type 2 diabetes mellitus (T2DM) patients feature a distinct gut microbiome signature4, while modulating the gut microbiome by either antibiotics or fecal microbial transplantation (FMT) is suggested to impact insulin sensitivity. Originally designed to treat obesity, bariatric surgeries often induce a robust and rapid weight-independent improvement in glucose homeostasis within days. Early diabetes remission following bariatric surgery is hypothesized to be mediated by rapid alterations in the gut microbiome and bile acids composition, however, the exact mechanism is yet to be uncovered. Elucidating this mechanism is important as it may form the basis of a new therapeutic modality in diabetes. The investigators intend to deeply characterize early post-bariatric changes in the gut microbiome of diabetic patients, as well as their gut mucosal transcriptome and metabolome, by using state-of-the-art experimental and computational pipelines. Additionally, The investigators will utilize a unique mouse model of bariatric surgery under germ-free conditions, developed at the Elinav lab, that allows us to dissect the role of microbes in post-operative metabolic improvements.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is one of the most prevalent and deadly conditions in the 21st century. T2DM is characterized by obesity and insulin resistance that leads to chronic hyperglycemia, which even with best medical care is often uncontrolled, resulting in life-threatening micro- and macrovascular complications.

The gut microbiota (i.e. the microbial population inhabiting the gut) has been extensively linked to blood glucose levels and was shown to mediate insulin response in various settings, including anti-diabetic pharmacotherapy. Moreover, fecal microbial transplantation (FMT) from lean healthy donors improved insulin resistance in humans suffering from metabolic syndrome. These pre-clinical and clinical evidence suggest that the gut microbiota has a mechanistic role in insulin-resistance.

Bariatric surgeries were originally designed to treat obesity but were also retrospectively found to ameliorate T2DM among other metabolic and non-metabolic disorders. Since obesity is a significant risk factor for T2DM, it is not surprising that surgically-induced weight loss which occurs within several months after surgery also improves insulin sensitivity. However, a substantial share of patients experience an improvement in insulin resistance within days after bariatric surgery, which clinically presents as normal glycemic values despite decreased dosage of anti-diabetic medications in the first post-operative days. This phenomenon of early diabetes remission after surgery precedes any weight-loss, therefore it is weight-independent and it is far from being understood.

Several explanations were suggested to explain early post-bariatric surgery diabetes remission, among which are acute caloric restriction, amplified incretins response, and rapid alterations in bile acids composition; however, none of them accounts for such a drastic improvement in glycemic control within such a short time frame.

Bariatric surgery rapidly alters the gut microbiome in a conserved fashion in both humans and rodents. Although descriptive studies demonstrated a change in microbiome composition within a few months after surgery, most studies didn't analyze microbiome in the first post-operative weeks in which the improvement in diabetes takes place, and data so far remains associative at best. Two independent studies exhibited improved metabolism following FMT from post-bariatric surgery humans and mice donors

into germ-free (microbiota-devoid) mice recipients, however, no mechanism was suggested and both studies used stool samples taken at a very late postoperative period, therefore no conclusions could be made regarding early diabetic remission. Caloric restriction, incretins, bile-acids, and the gut microbiome most probably "co-evolve" following surgery to exert surgery's beneficial metabolic effect with no single factor solely responsible for the entire effect.

Despite being highly effective in ameliorating obesity and obesity-related co-morbidities in the short-term, bariatric surgeries are invasive, risky, and not always successful in the long-term. Bariatric surgeries are thus far from being a perfect solution to obese diabetic patients, but they do serve as an intriguing investigational-model in the context of glucose metabolism. Hopefully, probing the mechanisms behind surgery's metabolic effect will facilitate the development of safer treatments for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult Population (> 18 years old)
* Diabetic Patients (Type 2)
* Bariatric surgery candidates for two types of bariatric surgery, i.e. sleeve gastrectomy and Roux-en-Y gastric bypass
* Laparoscopic Cholecystectomy candidates

Exclusion Criteria:

* Pregnant Women
* < 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in intestinal microbiota composition prior and following bariatric surgery | two weeks
  Changes in intestinal microbiota composition following bariatric surgery measured with RNA sequencing
Changes in glycemic index prior and following bariatric surgery | two weeks
  Changes in glycemic index prior and following bariatric surgery measured with continues glucose monitoring system (FreeStyle Libre)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Tel Aviv (Gosh Dan), Israel

IPD SHARING:
Plan to Share IPD: No